CLINICAL TRIAL: NCT04023448
Title: The Effect of Different Reconstruction Methods in Laparoscopic Anterior Rectal Resection on Postoperative Anterior Resection Syndrome：a Randomized Controlled Trial
Brief Title: The Effect of Different Reconstruction Methods on Anterior Resection Syndrome
Acronym: TEDRMARS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Hongbo Wei, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CPSCA-01
Record Dates: First submitted 2019-07-13; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Rectal Cancer; Low Anterior Resection Syndrome
Keywords: rectal cancer
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- coloplasty(CP) (Experimental): After purse-string suture and ligation of the head of the stapler at the colonic end, 5cm away from the colonic end, 5cm longitudinal incision was made to the proximal end of the teniae coli in the anterior wall of the colon, transverse suture was performed, and the plasmomuscular layer was embedded, then end to end colon-rectum (or anal canal) anastomosis was performed
  Interventions: Procedure: transverse coloplasty pouch
- straight colorectal anastomosis (SCA) (No Intervention): End to end colon-rectum (or anal canal) anastomosis was performed routinely

INTERVENTIONS:
Procedure: transverse coloplasty pouch — a transverse coloplasty pouch was performed before end to end colon-rectum (or anal canal) anastomosis
  Arms: coloplasty(CP)

SUMMARY:
The incidence of prerectal resection syndrome (LARS) after middle and low rectal cancer surgery is as high as 70%, which seriously affects the quality of life of patients. Studies have shown that colon pouch can reduce and alleviate LARS symptoms. However, most previous studies focused on open surgery, and the evaluation index lacked objectivity. Therefore, in the context of minimally invasive rectal cancer surgery, it is necessary to re-evaluate the value of improved surgical methods for the prevention of LARS, so as to improve the quality of life of patients.

DETAILED DESCRIPTION:
The incidence of prerectal resection syndrome (LARS) after middle and low rectal cancer surgery is as high as 70%, which seriously affects the quality of life of patients. LARS may be related to the injury of anal internal sphincter, anal sensory nerve injury, defecation reflex pathway injury, changes in anorectal Angle and rectum sigmoid Angle, changes in new rectal sensory function and compliance, and changes in dynamics,etc. After AR surgery, the rectum loses its good compliance and the storage capacity is reduced, which is one of the important reasons for the increased frequency and urgency of defecation.Therefore, on the basis of traditional colon-rectum (or anal canal) end-to-end anastomosis, "J" shaped pouch anastomosis, end-to-end anastomosis, coloplasty and other special anastomosis methods were performed. Meanwhile, for the lack of objective evaluation index, the results were not credible. The LARS score was first published in 2012,and has been validated, evaluated, or used as an outcome measure in more than 30 published scientific papers. Further more,laparoscopic surgery is widely used in gastrointestinal surgery. Herein, current randomized controlled trial comparing coloplasty with straight colorectal anastomosis in LARS in order to guide clinical practise was conducted.

ELIGIBILITY:
Inclusion Criteria:

* 20 years old ≤80 years old, regardless of gender, signed informed consent,
* BMI≤kg/m^2,
* Primary rectal lesions are pathologically diagnosed as rectal adenocarcinoma by endoscopic biopsy,
* The distance between the tumor and the anal margin is 5cm to 12cm,
* Preoperative tumor stage is T1-4N0-3M0,(according to AJCC-8th TNM tumor staging),
* Normal anorectal function and LARS score ≤20.

Exclusion Criteria:

* Patients with inflammatory bowel disease, chronic constipation, irritable bowel syndrome and other intestinal diseases that may affect bowel function,
* Patients with large tumors or extensive invasion of surrounding tissues and organs, TME is not applicable,
* Long-term use of drugs (such as morphine) that may affect bowel function,
* Patients with a history of abdominal, pelvic and anorectal surgery,
* Patients with severe mental illness or who cannot be evaluated due to cultural or psychological reasons.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
anterior resection syndrome incidence | 1 year after surgery
  LARS score≥21

SECONDARY OUTCOMES:
Early postoperative complication incidence | 30 days after surgery
  Anastomotic fistula, Hemorrhage, Pulmonary infection，Death
Length of hospital stay after surgery | 30 days after surgery
  Length of hospital stay
Bowel recovery time | 7 days after surgery
  Time interval from surgery to flatus and defecation
Long-term postoperative complication incidence | 1 year after surgery
  Anastomotic fistula, Hemorrhage，Intestinal obstruction

CONTACTS AND LOCATIONS:
Overall Officials: Hongbo Wei, Ph.D, Study Director — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-Sen university, Guanzhou, Guangdong, China